CLINICAL TRIAL: NCT06086054
Title: Effectiveness of a Childcare Intervention on Retention in the Cervical Cancer Screening and Diagnostic Continuum
Brief Title: Effect of a Childcare Resource on Cervical Cancer Prevention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Our previous childcare vendor's contract ended in January of 2025 and was not renewed. As of June 2025, a new vendor was still not established, and the decision was made by the study team to discontinue enrollment.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Robert Martin, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STU-2021-0309
Record Dates: First submitted 2023-09-14; First posted 2023-10-17 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Cervical Dysplasia
Keywords: Childcare; Social determinant of health; Patient navigation
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): The intervention is comprised of two components to link randomized patients to our health system childcare facility: 1) navigation by the research assistant to the childcare facility and 2) placement of the facility EMR referral. Navigation will occur an eligible patient is randomized to the intervention group. Navigation will consist of the research assistant educating the patient about the childcare facility and providing information about how to access the childcare facility during the telephone contact and via mailed written materials.
  Interventions: Behavioral: Navigation and EMR referral to childcare facility
- Standard Care (No Intervention): Patients randomized to the control group will undergo current standard of care with regards to childcare, which currently consists of passive sources of information about our childcare facility (Parkland website, signage in the hospital, or via word of mouth). Currently, there is no formalized mechanism for patients referred to gynecology from primary care to receive information about childcare aside from the above passive sources of information.

INTERVENTIONS:
Behavioral: Navigation and EMR referral to childcare facility — See arm description
  Arms: Intervention

SUMMARY:
Aim 1: Determine the prevalence of unmet childcare needs among women with abnormal cervical cancer screening and establish the relevance of childcare as a social determinant of health in the context of cervical dysplasia.

Aim 2: Conduct a pilot pragmatic patient-randomized control trial (RCT) to evaluate the effectiveness of an intervention linking eligible patients to our childcare facility compared to standard of care on retention in care, defined as show-rate for the initial visit in the gynecology dysplasia clinic. The intervention will consist of 1) patient navigation to our childcare facility prior to the initial visit in the gynecology dysplasia clinic and 2) placement of an electronic medical record (EMR) referral to our childcare facility.

Hypothesis: The study team hypothesizes that women receiving the intervention will have increased retention in care compared to women randomized to standard of care among women with abnormal cervical cancer screening referred to gynecology for diagnostic work-up.

These two aims will demonstrate the significance of childcare as a social determinant of health in the cervical cancer screening and diagnostic continuum by assessing the burden of unmet childcare needs among women with cervical dysplasia and measuring the effect of health system-integrated childcare as an intervention for unmet childcare needs on retention in care and subsequent completion of diagnostic work-up among women with cervical dysplasia. This study will rigorously provide the first evidence illustrating the effect of health systems' investment in addressing unmet childcare needs on preventive care like cervical cancer screening. The findings of this proposed pilot study will be utilized to develop future large-scale studies with extramural funding, building a longitudinal program of research on addressing childcare as a social determinant of health in this and other similar clinical contexts (e.g., breast cancer screening and treatment).

ELIGIBILITY:
Inclusion Criteria:

* All women with abnormal cervical cancer screening referred to Parkland gynecology dysplasia clinic as a new patient

Exclusion Criteria:

* Pregnant women
* Patients <18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Show-rate for initial visit to gynecology dysplasia clinic | Up to 2 years
  Show-rate assessed via EMR

SECONDARY OUTCOMES:
Rate of completion of indicated diagnostic and therapeutic procedures | Up to 2 years
  May include colposcopy, biopsies, and cervical excisional procedures, including hysterectomy, in the clinic and operating room (OR). Will vary based on clinical indication and assessment during initial appointment.
Show-rate for follow-up visits in gynecology | Up to 2 years
  Show-rate assessed via EMR
Rate of utilization of childcare facility during scheduled gynecology visits | Up to 2 years
  Rate of utilization assessed by health system's dashboard for childcare facility

OTHER OUTCOMES:
Questionnaire of patient-centered outcomes about experience in health system and in gynecology clinic | Up to 2 years
  Designed questions in a follow-up survey administered via telephone after initial appointment

CONTACTS AND LOCATIONS:
Overall Officials: Anisha Ganguly, MD, MPH, Principal Investigator — Parkland Health & Hospital System - - Dallas, TX
Locations (1):
- Parkland Health, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This is not permitted under our system's Office of Research Administration policies with regards to this type of collected patient data.

REFERENCES:
- [Background] Alvarez KS, Bhavan K, Mathew S, Johnson C, McCarthy A, Garcia B, Callies M, Stovall K, Harms M, Kho KA. Addressing childcare as a barrier to healthcare access through community partnerships in a large public health system. BMJ Open Qual. 2022 Oct;11(4):e001964. doi: 10.1136/bmjoq-2022-001964. PMID 36261213